CLINICAL TRIAL: NCT00356421
Title: A 52-Week Multicenter, Open-Label, Randomized, Parallel, Two - Arm Study Comparing Exubera® (Inhaled Human Insulin) Vs. Humalog® (Insulin Lispro), Both In Combination With Insulin Glargine In Subjects With Type 1 Diabetes Mellitus
Brief Title: A Clinical Trial Comparing Efficacy and Safety of Exubera® and Humalog®
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2171035
Record Dates: First submitted 2006-07-24; First posted 2006-07-26 (Estimated); Results first posted 2009-08-11 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-01

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Exubera; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Drug: Insulin lispro (Humalog)
- Experimental (Experimental)
  Interventions: Drug: Inhaled Human Insulin (Exubera®)

INTERVENTIONS:
Drug: Inhaled Human Insulin (Exubera®) — Preprandial inhaled insulin regimen and administration of insulin glargine QD
  Arms: Experimental
Drug: Insulin lispro (Humalog) — Subcutaneous insulin regimen of pre-prandial insulin lispro and administration of insulin glargine QD.
  Arms: Control

SUMMARY:
To compare efficacy and safety of Exubera® vs Humalog in patients with type 1 diabetes mellitus

DETAILED DESCRIPTION:
Pfizer announced in October 2007 that it would stop marketing Exubera®. At that time recruitment for study, A2171035 was placed on hold. Nektar, the company from which Pfizer licensed Exubera®, announced on April 9, 2008 that it had stopped its search for a new marketing partner. Accordingly, there will be no commercial availability of Exubera®. As a result, study A2171035 was terminated on May 12, 2008. Neither safety nor efficacy reasons were the cause of the study termination.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus Type 1

Exclusion Criteria:

* Severe Asthma, severe Chronic Obstructive Pulmonary Disease (COPD)
* Smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2006-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- United States (2):
  - Pfizer Investigational Site, Hamilton, New Jersey
  - Pfizer Investigational Site, New Brunswick, New Jersey
- Pfizer Investigational Site, Vienna, Austria
- Belgium (3):
  - Pfizer Investigational Site, Edegem
  - Pfizer Investigational Site, Genk
  - Pfizer Investigational Site, Leuven
- Pfizer Investigational Site, Aarhus, Denmark
- Pfizer Investigational Site, Kuopio, Finland
- France (3):
  - Pfizer Investigational Site, Brest
  - Pfizer Investigational Site, Corbeil-Essonnes
  - Pfizer Investigational Site, Strasbourg
- Pfizer Investigational Site, Waterford, Ireland
- Pfizer Investigational Site, Amsterdam, Netherlands
- Pfizer Investigational Site, Stavanger, Norway
- Pfizer Investigational Site, Lisbon, Portugal
- Spain (2):
  - Pfizer Investigational Site, Las Palmas, LAS Palmas de GRAN Canaria
  - Pfizer Investigational Site, Valencia, Valencia
- Pfizer Investigational Site, Stockholm, Sweden
- United Kingdom (3):
  - Pfizer Investigational Site, Bournemouth, Dorset
  - Pfizer Investigational Site, Dundee, Tayside
  - Pfizer Investigational Site, Birmingham, West Midlands

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171035&StudyName=A%20Clinical%20Trial%20Comparing%20Efficacy%20and%20Safety%20of%20Exubera%20and%20Humalog

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 340 subjects were planned to be randomized; 87 were screened and 58 were randomized to study treatment prior to study termination.
Pre-assignment Details: As a result of Pfizer's decision (18Oct2007) to return the worldwide rights for Exubera ® (insulin human [rDNA origin]) Inhalation Powder) to Nektar, from which Pfizer licensed inhaled insulin technology, it was decided to terminate this study.
Groups:
- Exubera ®: Preprandial inhaled insulin regimen plus once daily (QD) administration of insulin glargine.
- Insulin Lispro: Subcutaneous (SC) insulin regimen of pre-prandial insulin lispro and QD administration of insulin glargine.
Period: Overall Study
Arm/Group | Exubera ® | Insulin Lispro
Started | 38 | 20
Completed | 6 | 3
Not Completed | 32 | 17
Not completed — Lack of Efficacy | 3 | 0
Not completed — Withdrawal by Subject | 9 | 2
Not completed — Related to study drug | 15 | 12
Not completed — Not related to study drug | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exubera ® | Insulin Lispro | Total
Number analyzed (Participants) | 38 | 20 | 58
Age, Customized [Number; unit: participants] — Safety population.
  participants
    18 - 44 years | 22 | 13 | 35
    45 - 64 years | 14 | 6 | 20
    >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 6 | 23
  Male | 21 | 14 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) Percent (%)
Description: As a result of Pfizer's decision (18Oct2007) to return the worldwide rights for Exubera ® (insulin human [rDNA origin]) Inhalation Powder) to Nektar, from which Pfizer licensed inhaled insulin technology, it was decided to terminate this study. No efficacy data were summarized due to limited enrollment/early termination.
Time Frame: At 52 weeks
Population: Intent to Treat (ITT) population. Due to low number of subjects that completed, no descriptive statistics for the efficacy endpoints are provided.
Measure: Number; unit: percent
Arm/Group | Exubera ® | Insulin Lispro
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Subjects Who Attained HbA1c Levels of <8%, <7%, <6.5%, and >=8%
Description: as for outcome 1
Time Frame: At 52 weeks
Population: ITT population. Due to low number of subjects that completed, no descriptive statistics for the efficacy endpoints are provided.
Measure: Number; unit: percent
Arm/Group | Exubera ® | Insulin Lispro
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Subjects With Absolute Reduction in HbA1c Levels From Baseline of >0.5%, >0.7% and >1.0%
Description: as for outcome 1
Time Frame: At 52 weeks
Population: as for outcome 2
Measure: Number; unit: percent
Arm/Group | Exubera ® | Insulin Lispro
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Subjects Who Attained Target Fasting Plasma Glucose (FPG) Values (4.0 to 6.5 mmol/l; 72 to 117 mg/dl) From Baseline
Description: as for outcome 1
Time Frame: At weeks 2, 4, 6, 12, 24, 36, and 52 or last observation.
Population: as for outcome 2
Measure: Number; unit: percent
Arm/Group | Exubera ® | Insulin Lispro
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in FPG
Description: as for outcome 1
Time Frame: At 52 weeks or last observation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dl)
Arm/Group | Exubera ® | Insulin Lispro
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Fasting Blood Glucose Based on Glucometer Data and In-hospital Assessments
Description: as for outcome 1
Time Frame: To 52 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Exubera ® | Insulin Lispro
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Post-prandial Blood Glucose Based on Glucometer Data and In-hospital Assessments
Description: as for outcome 1
Time Frame: To 52 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Exubera ® | Insulin Lispro
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Insulin Antibody Levels
Description: as for outcome 1
Time Frame: At weeks 24 and 52 or last observation.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Exubera ® | Insulin Lispro
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline in Body Weight
Description: as for outcome 1
Time Frame: At weeks 12, 24, 36, and 52 or last observation.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Exubera ® | Insulin Lispro
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Body Mass Index
Description: as for outcome 1
Time Frame: At weeks 12, 24, 36, and 52 or last observation.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilograms per meter squared (kg/m2)
Arm/Group | Exubera ® | Insulin Lispro
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline in Basal Insulin Doses
Description: as for outcome 1
Time Frame: To 52 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: International Units (IU)
Arm/Group | Exubera ® | Insulin Lispro
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change From Baseline in Prandial Insulin Doses
Description: as for outcome 1
Time Frame: To 52 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Exubera ® | Insulin Lispro
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Blood Glucose Values From Baseline Determined by Home-monitored Blood Glucose (Subject Recorded Worksheet Values)
Description: as for outcome 1
Time Frame: To 52 weeks.
Population: as for outcome 2
Measure: Number; unit: mg/dl
Arm/Group | Exubera ® | Insulin Lispro
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: Subject Reported Health State From Baseline as Measured in the EuroQol-5 Dimensions (EQ-5D) Questionnaire
Description: as for outcome 1
Time Frame: At weeks 6, 24, and 52 or last observation
Population: as for outcome 2
Measure: Number; unit: scores on scale
Arm/Group | Exubera ® | Insulin Lispro
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Change in Fasting Lipids From Baseline
Description: as for outcome 1
Time Frame: At weeks 24 and 52 or last observation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Exubera ® | Insulin Lispro
Number analyzed (Participants) | 0 | 0

16. Other Pre Specified Outcome: Subject Reported Quality of Life From Baseline as Determined From Phase V System Measurement
Description: as for outcome 1
Time Frame: At weeks 6, 24, and 52 or last observation
Population: as for outcome 2
Measure: Number; unit: scores on scale
Arm/Group | Exubera ® | Insulin Lispro
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Exubera ® | Insulin Lispro
Serious Adverse Events (participants affected / at risk) | 2 | 1
Other Adverse Events (participants affected / at risk) | 35 | 20
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Exubera ® | Insulin Lispro
Blood creatinine increased (Investigations) | 1/38 | 0/20
Hypoglycaemia (Metabolism and nutrition disorders) | 2/38 | 0/20
Ketoacidosis (Metabolism and nutrition disorders) | 1/38 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Exubera ® | Insulin Lispro
Lymphadenitis (Blood and lymphatic system disorders) | 0/38 | 1/20
Vertigo (Ear and labyrinth disorders) | 1/38 | 0/20
Abdominal pain (Gastrointestinal disorders) | 0/38 | 1/20
Aphthous stomatitis (Gastrointestinal disorders) | 1/38 | 0/20
Dyspepsia (Gastrointestinal disorders) | 1/38 | 0/20
Haemorrhoids (Gastrointestinal disorders) | 0/38 | 1/20
Nausea (Gastrointestinal disorders) | 2/38 | 1/20
Vomiting (Gastrointestinal disorders) | 3/38 | 2/20
Asthenia (General disorders) | 1/38 | 0/20
Chest pain (General disorders) | 0/38 | 1/20
Drug intolerance (General disorders) | 1/38 | 0/20
Fatigue (General disorders) | 0/38 | 1/20
Hunger (General disorders) | 2/38 | 0/20
Malaise (General disorders) | 2/38 | 0/20
Pyrexia (General disorders) | 0/38 | 1/20
Balanitis candida (Infections and infestations) | 0/38 | 1/20
Ear infection (Infections and infestations) | 1/38 | 0/20
Gastroenteritis (Infections and infestations) | 3/38 | 1/20
Gastrointestinal infection (Infections and infestations) | 1/38 | 0/20
Influenza (Infections and infestations) | 2/38 | 1/20
Localised infection (Infections and infestations) | 2/38 | 0/20
Nasopharyngitis (Infections and infestations) | 9/38 | 7/20
Onychomycosis (Infections and infestations) | 1/38 | 0/20
Pharyngitis (Infections and infestations) | 0/38 | 2/20
Respiratory tract infection (Infections and infestations) | 0/38 | 2/20
Respiratory tract infection viral (Infections and infestations) | 1/38 | 0/20
Sinusitis (Infections and infestations) | 2/38 | 0/20
Tooth abscess (Infections and infestations) | 0/38 | 1/20
Tracheitis (Infections and infestations) | 1/38 | 0/20
Upper respiratory tract infection (Infections and infestations) | 0/38 | 1/20
Vaginal candidiasis (Infections and infestations) | 1/38 | 0/20
Viral pharyngitis (Infections and infestations) | 1/38 | 0/20
Vulvovaginitis (Infections and infestations) | 1/38 | 0/20
Eye injury (Injury, poisoning and procedural complications) | 1/38 | 0/20
Fall (Injury, poisoning and procedural complications) | 1/38 | 0/20
Joint sprain (Injury, poisoning and procedural complications) | 0/38 | 1/20
Thermal burn (Injury, poisoning and procedural complications) | 1/38 | 0/20
Wound (Injury, poisoning and procedural complications) | 1/38 | 0/20
Alanine aminotransferase increased (Investigations) | 1/38 | 0/20
Weight decreased (Investigations) | 1/38 | 0/20
Weight increased (Investigations) | 1/38 | 0/20
Anorexia (Metabolism and nutrition disorders) | 1/38 | 0/20
Hyperglycaemia (Metabolism and nutrition disorders) | 2/38 | 1/20
Hypoglycaemia (Metabolism and nutrition disorders) | 33/38 | 18/20
Polydipsia (Metabolism and nutrition disorders) | 1/38 | 0/20
Arthralgia (Musculoskeletal and connective tissue disorders) | 2/38 | 0/20
Back pain (Musculoskeletal and connective tissue disorders) | 2/38 | 1/20
Bone pain (Musculoskeletal and connective tissue disorders) | 1/38 | 0/20
Joint swelling (Musculoskeletal and connective tissue disorders) | 1/38 | 0/20
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0/38 | 1/20
Myalgia (Musculoskeletal and connective tissue disorders) | 1/38 | 0/20
Myositis (Musculoskeletal and connective tissue disorders) | 1/38 | 0/20
Neck pain (Musculoskeletal and connective tissue disorders) | 1/38 | 0/20
Tendonitis (Musculoskeletal and connective tissue disorders) | 1/38 | 0/20
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/38 | 1/20
Disturbance in attention (Nervous system disorders) | 1/38 | 0/20
Dizziness (Nervous system disorders) | 2/38 | 0/20
Headache (Nervous system disorders) | 4/38 | 1/20
Somnolence (Nervous system disorders) | 1/38 | 0/20
Tremor (Nervous system disorders) | 1/38 | 0/20
Depression (Psychiatric disorders) | 1/38 | 0/20
Disorientation (Psychiatric disorders) | 1/38 | 0/20
Mental disorder (Psychiatric disorders) | 1/38 | 0/20
Ketonuria (Renal and urinary disorders) | 0/38 | 1/20
Polyuria (Renal and urinary disorders) | 1/38 | 0/20
Endometriosis (Reproductive system and breast disorders) | 1/38 | 0/20
Cough (Respiratory, thoracic and mediastinal disorders) | 5/38 | 0/20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/38 | 0/20
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0/38 | 1/20
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1/38 | 0/20
Pharyngolaryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0/38 | 1/20
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2/38 | 2/20
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0/38 | 1/20
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2/38 | 0/20
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 4/38 | 0/20
Pruritus (Skin and subcutaneous tissue disorders) | 1/38 | 0/20
Rash macular (Skin and subcutaneous tissue disorders) | 0/38 | 1/20
Haematoma (Vascular disorders) | 1/38 | 1/20
Hot flush (Vascular disorders) | 1/38 | 0/20
Hypertensive crisis (Vascular disorders) | 1/38 | 0/20

LIMITATIONS AND CAVEATS:
As a result of Pfizer's decision to stop marketing Exubera ®, this study was terminated. Due to the early termination of the study and the low number of subjects who completed, no descriptive statistics for efficacy endpoints are provided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.